CLINICAL TRIAL: NCT00441584
Title: Efficacy and Safety of PEG-Intron Plus Rebetol in Subjects With Chronic Hepatitis C Genotype 1 Non Responder to Pegasys
Brief Title: The Effects of PegIntron Plus Rebetol in Subjects With Chronic Hepatitis C Not Responding to Pegasys (Study P03833)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Subject accrual was prematurely terminated due slow enrollment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03833; ESPECIAL
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PegIntron plus Rebetol (Experimental): PegIntron 1.5 μg/kg/week plus Rebetol 800-1400 mg/day administered for 48 weeks
  Interventions: Biological: PegIntron (peginterferon alfa-2b); Drug: Rebetol (ribavirin)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b) — Powder for injection in vial or Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  Other Names: SCH 54031, PEG-Intron, PegIntron, ViraferonPeg, peginterferon alfa-2b
Drug: Rebetol (ribavirin) — 200 mg capsules, oral, weight based dose of 800-1400 mg, daily for up to 48 weeks
  Other Names: SCH 18908, Rebetol, REBETOL, ribavirin

SUMMARY:
This is an uncontrolled, non-randomized, open-label, multinational study designed to evaluate the efficacy and safety of PegIntron plus Rebetol in subjects with chronic hepatitis C. The study is designed to determine the proportion of chronic hepatitis C genotype 1 subjects who did not respond to previous treatment with Pegasys 180µg QW plus ribavirin, that will achieve sustained virological response (SVR) when treated with PegIntron plus Rebetol.

ELIGIBILITY:
Inclusion Criteria:

* Subject must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subject must be 18-70 years of age of either sex and of any race.
* Subject must be diagnosed with chronic hepatitis C genotype 1 (confirmation by biopsy not required). (Liver function tests (LFTs) can be normal or elevated.)
* Female subjects cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile or using 2 methods of birth control. While abstinence from sexual activity is the only certain method to prevent pregnancy, female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use a combination of the following 2 methods:

  * Contraceptive pill or intrauterine device (IUD) or depot hormonal preparation (ring, injection, implant), and
  * A barrier method of contraception such as diaphragm, sponge with spermicide, condom, or a method of birth control considered acceptable by the study physician.
* Contraceptive measures will be reviewed with female subjects at each visit. Dual methods of contraception must be used for 6 months after treatment discontinuation.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screen phase and during the study.
* Confirmation by the principal investigator or a sub-investigator that sexually active male subjects are practicing a method of contraception considered acceptable (vasectomy, condom plus spermicide, plus relationship with a female partner who practices an acceptable method of contraception). Contraception must be used during the treatment period and for seven months after the completion of therapy, including condom use by male subjects with pregnant partners.
* Subject must be free of any clinically significant disease that would interfere with study evaluations.
* Subject must understand, be able to and agree to adhere to the dosing and visit schedules.
* Compensated liver disease with the following minimum hematologic and biochemical criteria at the Day 1 visit within normal limits:

  * Hemoglobin values equal to or greater than 12 g/dL for females and 13 g/dL for males
  * White blood cell (WBC) count equal to or greater than 3,000/cu mm
  * Neutrophil count equal to or greater than 1,500/cu mm
  * Platelet count equal to or greater than 80,000/cu mm
  * Direct bilirubin within normal limits
  * Indirect bilirubin within normal limits (unless non-hepatitis related factors such as Gilbert's disease explain an indirect bilirubin rise). In such cases indirect bilirubin should be less than or equal to 3.0 mg/dL (less than or equal to 51.3 µmol/L)
  * Albumin within normal limits
  * Serum creatinine within normal limits
  * Subject must be a non-responder, defined as having received and not having responded to a prior treatment consisting of one course of Pegasys 180 mcg QW in combination with ribavirin 1000-1200 mg daily, with or without amantadine, for a minimum of 12 weeks and:

    * Subject must be found to be hepatitis C virus (HCV)-ribonucleic acid (RNA) positive with less than a 2-log drop at 12 weeks of treatment, or
    * is polymerase chain reaction (PCR)-positive at End Of Treatment, whether End Of Treatment happened at week 48 or earlier
* Subject must be off Pegasys/ribavirin at least 12 weeks prior to screen.
* Subject must have had no other treatment with any interferon except Pegasys.
* Subject must neither have received nor currently be on any other treatment for his chronic hepatitis C disease, except for amantadine.
* When available, historical liver biopsy with pathology report of the subject must confirm that the histological diagnosis is consistent with chronic hepatitis C.
* Subject must have a value of thyroid stimulating hormone within normal limits (whether euthyroid or requiring thyroid medications).
* Antinuclear antibodies must be less than or equal to 1:320.
* If abdominal imaging has been performed within 1 year prior to screen, it must not show evidence of focal mass suggestive of hepatoma and/or ascites.
* For subjects with a history of diabetes or hypertension, clearance from an ophthalmologist has to be obtained prior to treatment start.

Exclusion Criteria:

* Subject is a female who is pregnant or breastfeeding, or who intends to become pregnant during the study.
* Subject has used any investigational product within 30 days prior to enrollment or is currently involved in another clinical trial.
* Subjects weighing over 125 kg.
* Subject has any of the following causes for the liver disease based on subject history or biopsy (where applicable) other than chronic hepatitis C, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Non-alcoholic steatohepatitis (NASH)
  * Drug-related liver disease
* Subject has any clinically significant deviation from normal in the physical examination, chest x-ray, or electrocardiogram (ECG) that, in the investigator's judgment, may interfere with the study evaluation or affect subject safety.
* Subject is in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subject is part of the staff or a family member of the staff personnel directly involved with this study.
* Subject is a previously untreated subject.
* Subject has been treated with Pegasys + less than 1000 mg of ribavirin (instead of with 1000-1200 mg of ribavirin).
* Subject has been discontinued from Pegasys treatment at any week due to an adverse event.
* Subject is co-infected with human immunodeficiency virus (HIV) and/or hepatitis B virus (HBV).
* Subject is suspected to be hypersensitive to interferon alpha or Peg-Intron or ribavirin.
* Subject has previously received interferon, (except for the Pegasys flat dose 180 mcg QW for at least 12 weeks), thymosin or Cell Cept treatment or any other drug intended to treat chronic hepatitis C.
* Subject has had organ transplants other than cornea and hair transplant.
* Subject has a history of hepatocellular carcinoma or any other malignancy (except basal cell carcinoma) within the last 5 years or a suspected diagnosis of hepatocellular carcinoma or other malignancy, or an active malignancy.
* Known coagulation diseases such as hemophilia; hemoglobin diseases (e.g. thalassemia).
* Subject has glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Subject has an evidence of decompensated liver disease such as history or presence of ascites, bleeding varices, spontaneous encephalopathy.
* Subject has any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study as followed below:

  * Preexisting psychiatric condition, especially moderate to severe depression, or a history of severe psychiatric disorder, such as psychosis, suicidal ideation, or suicide attempts. Severe depression includes the following:

    * Hospitalization for depression
    * Electroconvulsive therapy for depression, or
    * Depression causing a prolonged absence from work or significantly altering daily functions.
* Subjects with mild depression may be considered for entry into the study provided that a pre-treatment assessment demonstrates that the subject's emotional status is clinically stable, in which case a management plan must be formulated for the subject; this management plan will become a part of the subject's medical record.

  * Craniocerebral trauma, which is not a concussion, or active seizure disorders requiring medication.
  * Clinically significant ECG abnormalities and/or cardiovascular dysfunction within 6 previous months (e.g., angina, congestive heart failure, recent myocardial infarction, or significant arrhythmia).
  * Chronic lung disease (e.g., chronic obstructive lung disease)
  * Poorly controlled diabetes mellitus: HbA1C more than or equal to 8.5%
  * Immune-mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis)
  * Clinical gout
  * Creatinine clearance less than or equal to 50 mL/min
  * any medical condition which may require use of chronic systemic steroids
* Subject is or was a substance abuser, such as alcohol (80 g/day or more), methadone, intravenous (IV), oral or inhaled drugs. To be considered for inclusion, the subject must have abstained and agree to abstain from using any of the above for at least 6 months. Subjects treated with buprenorphine (Subutex) who have been stable for 6 months may be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The majority of subjects who discontinued due to treatment failure were withdrawn from the study as non-responders according to protocol requirements.
Period: Overall Study
Arm/Group | PegIntron Plus Rebetol
Started | 117
Completed | 12
Not Completed | 105
Not completed — Lack of Efficacy | 79
Not completed — Withdrawal by Subject | 8
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 4
Not completed — Failure to meet eligibility criteria | 3

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.54 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Have Achieved Sustained Virological Response (SVR) at 24 Weeks Post End of Treatment
Description: Sustained virologic response is defined as a plasma HCV RNA level below Lower Level of Quantitation at 24 weeks post-treatment, which is < 30 IU/mL in this study.
Time Frame: Up to 48 weeks of treatment plus 24 weeks follow up
Population: The All Treated population included all subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 117
Participants | 1

ADVERSE EVENTS:
Arm/Group | PegIntron Plus REBETOL
Serious Adverse Events (participants affected / at risk) | 6/117
Other Adverse Events (participants affected / at risk) | 105/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Plus REBETOL (N=117)
MENINGITIS ASEPTIC (Infections and infestations) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
INTENTION TREMOR (Nervous system disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
PSEUDODEMENTIA (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Plus REBETOL (N=117)
LEUKOPENIA (Blood and lymphatic system disorders) | 8 (8)
NEUTROPENIA (Blood and lymphatic system disorders) | 12 (16)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (6)
DIARRHOEA (Gastrointestinal disorders) | 7 (8)
NAUSEA (Gastrointestinal disorders) | 17 (20)
ASTHENIA (General disorders) | 29 (40)
CHILLS (General disorders) | 13 (15)
FATIGUE (General disorders) | 33 (37)
INFLUENZA LIKE ILLNESS (General disorders) | 25 (86)
INJECTION SITE ERYTHEMA (General disorders) | 13 (13)
INJECTION SITE REACTION (General disorders) | 10 (25)
IRRITABILITY (General disorders) | 9 (9)
PYREXIA (General disorders) | 23 (32)
INFLUENZA (Infections and infestations) | 17 (18)
NEUTROPHIL COUNT DECREASED (Investigations) | 7 (7)
ANOREXIA (Metabolism and nutrition disorders) | 14 (15)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 (21)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 (20)
DIZZINESS (Nervous system disorders) | 7 (7)
HEADACHE (Nervous system disorders) | 29 (31)
DEPRESSION (Psychiatric disorders) | 10 (11)
INSOMNIA (Psychiatric disorders) | 8 (10)
SLEEP DISORDER (Psychiatric disorders) | 12 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 (25)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 (11)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 11 (11)
ECZEMA (Skin and subcutaneous tissue disorders) | 7 (8)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 8 (8)
PRURITUS (Skin and subcutaneous tissue disorders) | 18 (18)

LIMITATIONS AND CAVEATS:
Due to slow enrollment, an unplanned interim analysis was conducted: 75 of 93 (80.6%) subjects who had reached treatment Week 12 did not achieve early virologic response. Given the low likelihood of response, a decision was made to stop enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less